CLINICAL TRIAL: NCT07306403
Title: THE COMPARISON OF GELATIN SPONGE TO SUTURE ALONE ON POST OPERATIVE SWELLING AFTER EXTRACTION OF IMPACTED MANDIBULAR THIRD MOLAR.
Acronym: Gelatin Sponge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Watim Medical & Dental College (Other)
Responsible Party: Principal Investigator, Dr.Mohammad Irfan, The Comparison of Gelatin Sponge To Suture Alone on Post Operative Swelling After Extraction of Impacted Mandibular Third Molar, Watim Medical & Dental College
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: Ethical Review Board
Record Dates: First submitted 2025-11-28; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2024-08

CONDITIONS: Post Operative Swelling; Impacted Mandibular Third Molar Extraction
MeSH Terms: interventions — Sutures; Mitochondrial Swelling

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Gelatin Sponge (Other): Swelling
  Interventions: Device: Gelatin Sponge Sheet; Procedure: Swelling
- Suture Alone (Other): Swelling
  Interventions: Device: Gelatin Sponge Sheet; Procedure: Swelling

INTERVENTIONS:
Device: Gelatin Sponge Sheet — Gelatin sponge vs Suture Alone
  Other Names: Sponge Stone; Suture
Procedure: Swelling — Suture

SUMMARY:
This Study is designed for purpose to increase patient safety and reduce complications which occurs after mandibular 3rd molar extraction which is will increase discomfort after extraction. My study hypothesis is that gelatin sponge after extraction reduce swelling post extraction wisdom tooth.For understanding when we remove wisdom tooth, we involve hard and soft tissiues which will result in post extraction swelling.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-30 years old.
2. Either gender.
3. impacted third mandibular molar.
4. No history of periodontists
5. No bone recession on radiograph
6. Swelling at the side of impaction.

Exclusion Criteria:

1. Patients with ASA status lll and above.
2. -Patients requiring multiple extractions in same appointment.
3. Patients allergic to Lignocaine.
4. Patients in whom adrenaline is contraindicated.
5. Medically compromised individual such as those with poorly controlled diabetes, hypertension and pregnancy,

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Post Extraction Swelling | Pre extraction, 1st day post extraction, 3rd day post extraction and 7th day post extraction.
  Measurements will be taken from angle of mandible to commissure of lips by measuring tape by Amin and Laskin Method.

CONTACTS AND LOCATIONS:
Locations (1):
- Watim Medical and Dental College, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No
Because want to avoid sharing their identity